CLINICAL TRIAL: NCT03879837
Title: A Randomized, Blinded, Parallel Group, Placebo-Controlled, Multiple Dose, Multicenter Study to Compare the Therapeutic Equivalence of Fluticasone Propionate Pressurized Metered Dose Inhaler, 110 mcg, to Flovent® HFA 110 mcg, in Adult Subjects With Asthma
Brief Title: Therapeutic Equivalence of Fluticasone Propionate Pressurized Metered Dose Inhaler, 110 mcg, to Flovent® HFA 110 mcg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPI-18-03
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Asthma
Keywords: Bioequivalence
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Investigational Test Product (Experimental): Fluticasone propionate pressurized metered dose inhaler, 110 mcg per actuation
  Interventions: Drug: Fluticasone propionate pressurized metered dose inhaler
- Reference Listed Drug (Active Comparator): Flovent HFA pressurized metered dose inhaler, 110 mcg per actuation
  Interventions: Drug: Flovent HFA pressurized metered dose inhaler
- Placebo (Placebo Comparator): Placebo pressurized metered dose inhaler, no active content
  Interventions: Drug: Placebo pressurized metered dose inhaler

INTERVENTIONS:
Drug: Fluticasone propionate pressurized metered dose inhaler — 110 mcg per actuation
  Arms: Investigational Test Product
Drug: Flovent HFA pressurized metered dose inhaler — 110 mcg per actuation
  Other Names: Fluticasone propionate pressurized metered dose inhaler
  Arms: Reference Listed Drug
Drug: Placebo pressurized metered dose inhaler — no active content
  Arms: Placebo

SUMMARY:
A Randomized, Blinded, Parallel Group, Placebo-Controlled, Multiple Dose, Multicenter Study to Compare the Therapeutic Equivalence of Fluticasone Propionate Pressurized Metered Dose Inhaler, 110 mcg, to Flovent® HFA 110 mcg, in Adult Subjects with Asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥18 and ≤75 years of age male or female subjects of non-child bearing potential or of child bearing potential committing to consistent and correct use of an acceptable method of birth control.
2. Body mass index (BMI) ≥18 and ≤45.
3. Diagnosis of asthma, as defined by the NAEPP-EPR3 at least 12 months prior to Enrollment at Screening Visit 1a.
4. Pre bronchodilator highest forced expiratory volume in 1 second (FEV1) ≥45% and ≤85% of predicted normal value at Screening Visit 1b and on the first day of treatment prior to randomization.
5. Reversibility of airway obstruction ≥15% of FEV1 within 30 minutes of 360mcg albuterol inhalation (4 puffs).
6. Subjects should be stable on their chronic asthma treatment regimen for at least 4 weeks prior to Enrollment at Screening Visit 1a.
7. Currently non-smoking, defined as abstinence from all smoking, including marijuana and all tobacco products (i.e., e-cigarettes, cigarettes, cigars, pipe, ortobacco) within the past year, a negative cotinine screening test at Screening Visit 1b, and <10 pack years of historical use.
8. Able to replace current short-acting β agonist (SABA) with study issued albuterol inhaler for use as needed for the duration of the study.
9. Able to withhold all inhaled SABAs for at least 6 hours prior to lung function assessments on study visits.
10. Able to withhold all inhaled long acting β agonists (LABA) 24 hours before Screening Visit 1b.
11. Able to discontinue current asthma medications (e.g., inhaled corticosteroids[ICS], LABA, etc.) during the Run-in period and for remainder of the study.
12. Able to comply with study procedures, including correct use of inhaler devices and home peak expiratory flow (PEF) device, and maintaining an electronic diary (eDiary).
13. Willingness to give their written informed consent to participate in the study.

Exclusion Criteria:

1. Life-threatening asthma, defined as a history of asthma episodes(s) requiring intubation, and/or associated with hypercapnia, respiratory arrest or hypoxic seizures, asthma related syncopal episode(s), or hospitalizations due to asthma within the past year prior to Enrollment, or during the Screening or Run-in period.
2. History of significant respiratory disease other than asthma (e.g., chronic obstructive pulmonary disease [COPD], interstitial lung disease, chronic bronchitis, emphysema, etc.).
3. Evidence or history of clinically significant disease or abnormality including congestive heart failure, uncontrolled hypertension, uncontrolled coronary artery disease, myocardial infarction, or cardiac dysrhythmia. In addition, historical or current evidence of significant hematologic, hepatic, neurologic, psychiatric, renal, cardiovascular, endocrine, or other diseases that, in the opinion of the Investigator, would put the subject at risk through study participation, or would affect the study analyses if the disease exacerbates during the study.
4. Viral or bacterial, upper/lower respiratory tract infection (U/LRTI), or sinus, or middle ear infection within 4 weeks prior to Screening Visit 1b, during the Run-in period, or on the first day of treatment prior to randomization.
5. Hypersensitivity to any sympathomimetic drug (e.g., albuterol) or any inhaled, intranasal, or systemic corticosteroid therapy.
6. Hypersensitivity to any of the ingredients of FP pMDI or Flovent HFA.
7. Subjects receiving β2 blockers, anti-arrhythmics, anti-depressants, and/or monoamine oxidase inhibitors within 4 weeks prior to Screening Visit 1b.
8. Subjects who required systemic or oral corticosteroids (for any reason) within the past 6 months prior to Screening Visit 1b.
9. Subjects receiving medications that are strong cytochrome P4503A4 inhibitors (e.g., ritonavir, ketoconazole, itraconazole) within 2 weeks prior to Screening Visit 1b.
10. Subjects receiving any approved or investigational biological treatment for asthma (e.g., omalizumab, mepolizumab) within 6 months prior to Screening Visit 1b.
11. Subjects with clinically relevant abnormal chemistry laboratory findings at Screening Visit 1b as assessed by the Investigator.
12. Subjects with clinically significant electrocardiogram (ECG) findings at Screening Visit 1b as assessed by the Investigator and/or cardiologist.
13. Subjects who have received any Investigational Product (IP) within 1 month prior to Screening Visit 1b and as described in the Washout Table in Appendix 1.
14. Female subjects who are pregnant or breast feeding.
15. Evidence of oral candidiasis at Screening or randomization, or history within 1year prior to Screening Visit 1b.
16. Evidence or history of tuberculosis, hypercorticism, or adrenal suppression.
17. Evidence or history within the 6 months prior to Screening Visit 1b of clinically relevant eye problems such as cataracts. Any previous diagnosis or treatment for ocular hypertension or glaucoma is exclusionary.
18. Subjects with hyperbilirubinemia (defined as aspartate aminotransferase [AST] or alanine aminotransferase [ALT] ≥3 times the upper limit of the normal range [ULN], or bilirubin ≥2 times the ULN) or Hy's Law events.
19. Evidence or history of drug or alcohol abuse in the 2 years prior to Enrollment at Screening Visit 1a or a positive drug or alcohol test at Screening Visit 1b.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1902 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Mean change in baseline adjusted morning pre-dose FEV1 from the time of treatment randomization to Week 4. | 4 weeks

SECONDARY OUTCOMES:
Superiority over Placebo | Approximately 4 Weeks
  To confirm the Test and Reference listed Drug products are statistically superior to placebo (p< 0.05) on the primary study endpoint.

CONTACTS AND LOCATIONS:
Locations (1):
- Site 1, Spartanburg, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared.